CLINICAL TRIAL: NCT01095562
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Phase 2 Study of the Safety and Efficacy of ABT-126 in the Treatment of Cognitive Deficits in Schizophrenia (CDS)
Brief Title: Safety and Efficacy Study for Cognitive Deficits in Adult Subjects With Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M10-854
Record Dates: First submitted 2010-03-26; First posted 2010-03-30 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2013-01

CONDITIONS: Cognitive Deficits in Schizophrenia
MeSH Terms: interventions — ABT-126

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ABT-126 Dose 1 (Experimental)
  Interventions: Drug: ABT-126
- ABT-126 Dose 2 (Experimental)
  Interventions: Drug: ABT-126
- Sugar Pill (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ABT-126 — ABT-126 Dose 1, ABT-126 Dose 2
  Arms: ABT-126 Dose 1; ABT-126 Dose 2
Drug: Placebo — Placebo
  Arms: Sugar Pill

SUMMARY:
This is an efficacy and safety study evaluating an experimental treatment for cognitive deficits in adults with schizophrenia.

DETAILED DESCRIPTION:
This is a Phase 2 study designed to evaluate the efficacy and safety of ABT-126 in approximately 210 adults with schizophrenia. Subjects will be randomized to one of three treatment groups (ABT-126 Dose 1, ABT-126 Dose 2 or placebo) for a 12-week Treatment Period. The purpose of this research study is to find out whether ABT-126 compared to placebo can improve cognition and what side effects ABT-126 may cause. Cognition is the way a person thinks, and it includes abilities like paying attention, focusing, remembering things, and solving problems. Acronyms listed in the Outcomes and/or Eligibility sections for this study are defined below: • MCCB: Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery • UPSA-2: University of California at San Diego (UCSD) Performance-Based Skills Assessment-2 • CANTAB: Cambridge Neuropsychological Test Automated Battery • PANSS: Positive and Negative Syndrome Scale • NSA-16: Negative Symptom Assessment-16 • CGI-S: Clinical Global Impression - Severity

ELIGIBILITY:
Inclusion Criteria

* Has current DSM-IV-TR diagnosis of schizophrenia confirmed by the Mini-International Neuropsychiatric Interview.
* Is clinically stable while receiving antipsychotic therapy with one or two atypical antipsychotic medications: lack of hospitalizations from 4 months of Initial Screening Visit; taking same antipsychotic medication(s) for at least 8 weeks prior to the Day -1 visit; core positive symptoms of PANSS no worse than moderate in severity throughout Screening Period of at least 4 weeks.
* Has been diagnosed with or treated for schizophrenia for at least 2 years prior to Initial Screening Visit.
* Has had continuity in psychiatric care (e.g., mental health system, clinic or physician) for at least 6 months prior to Initial Screening Visit.
* Has an identified responsible contact person (e.g., family member, social worker, case worker, or nurse) that can provide support to the subject and ensure compliance with protocol requirements.

Exclusion Criteria

* Has valid current or past diagnosis of schizoaffective disorder, bipolar disorder, manic episode, dementia, posttraumatic stress disorder, obsessive compulsive disorder, or a current major depressive episode.
* Has history of substance abuse (excluding nicotine or tobacco products) or alcohol abuse within 6 months prior to Screening Visit; has a substance dependence disorder (excluding nicotine or tobacco products) that has not been remitted for at least 1 year prior to Initial Screening Visit.
* Is taking any medication for extrapyramidal symptoms at any time from the Initial Screening Visit until the Day -1 Visit.
* Is taking any antidepressant that is excluded, including tricyclic antidepressants and monoamine oxidase inhibitors, at any time from 8 weeks prior to the Day -1 Visit.
* Has significant suicidal ideation at Initial Screening Visit.
* Has had a suicide attempt within 1 year prior to the Day -1 Visit.
* Has participated in another trial utilizing the MATRICS Consensus Cognitive Battery (MCCB) or UCSD Performance-Based Skills Assessment (UPSA) (any version) within 6 months prior to Initial Screening Visit.
* Is currently enrolled in any form of cognitive remediation training.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 207 (Actual)
Dates: Start 2010-03; Primary Completion 2011-08 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Cognition: MCCB | Measurements from screening period through 12-week treatment period

SECONDARY OUTCOMES:
Functioning: UPSA-2 | Measurements from screening period through 12-week treatment period
Cognition: CANTAB | Measurements from screening period through 12-week treatment period
Symptom Severity: PANSS, NSA-16, CGI-S | Measurements from screening period through 12-week treatment period

CONTACTS AND LOCATIONS:
Overall Officials: George Haig, PharmD, Study Director — AbbVie
Locations (23):
- United States (23):
  - Site Reference ID/Investigator# 26267, Cerritos, California
  - Site Reference ID/Investigator# 45320, Costa Mesa, California
  - Site Reference ID/Investigator# 27068, Escondido, California
  - Site Reference ID/Investigator# 52568, Garden Grove, California
  - Site Reference ID/Investigator# 26266, Granada Hills, California
  - Site Reference ID/Investigator# 26388, Oceanside, California
  - Site Reference ID/Investigator# 45315, San Bernardino, California
  - Site Reference ID/Investigator# 26271, San Diego, California
  - Site Reference ID/Investigator# 27045, Santa Ana, California
  - Site Reference ID/Investigator# 45314, Santa Ana, California
  - Site Reference ID/Investigator# 26264, Torrance, California
  - Site Reference ID/Investigator# 27072, Tampa, Florida
  - Site Reference ID/Investigator# 27043, Wichita, Kansas
  - Site Reference ID/Investigator# 26395, Lake Charles, Louisiana
  - Site Reference ID/Investigator# 26268, St Louis, Missouri
  - Site Reference ID/Investigator# 26392, Fresh Meadows, New York
  - Site Reference ID/Investigator# 27073, New York, New York
  - Site Reference ID/Investigator# 26262, Rochester, New York
  - Site Reference ID/Investigator# 27071, Beachwood, Ohio
  - Site Reference ID/Investigator# 36020, Media, Pennsylvania
  - Site Reference ID/Investigator# 28063, Norristown, Pennsylvania
  - Site Reference ID/Investigator# 27070, Sellersville, Pennsylvania
  - Site Reference ID/Investigator# 27069, Dallas, Texas

REFERENCES:
- [Background] Hashimoto K. Targeting of alpha7 Nicotinic Acetylcholine Receptors in the Treatment of Schizophrenia and the Use of Auditory Sensory Gating as a Translational Biomarker. Curr Pharm Des. 2015;21(26):3797-806. doi: 10.2174/1381612821666150605111345. PMID 26044974
- [Derived] Georgiades A, Davis VG, Atkins AS, Khan A, Walker TW, Loebel A, Haig G, Hilt DC, Dunayevich E, Umbricht D, Sand M, Keefe RSE. Psychometric characteristics of the MATRICS Consensus Cognitive Battery in a large pooled cohort of stable schizophrenia patients. Schizophr Res. 2017 Dec;190:172-179. doi: 10.1016/j.schres.2017.03.040. Epub 2017 Apr 20. PMID 28433500